CLINICAL TRIAL: NCT02495532
Title: Randomized Clinical Trial Comparing Carnoy's and GEWF Solutions for Lymph Node Clearing Technique in Colorectal Cancer
Brief Title: Clinical Trial Comparing Carnoy's and GEWF Solutions for Lymph Node Clearing Technique in Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Moinhos de Vento (Other)
Collaborators: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 39919814.7.0000.5330
Record Dates: First submitted 2015-04-16; First posted 2015-07-13 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Colorectal Neoplasms; Neoplasm Metastasis
Keywords: Neoplasm Metastasis; Colorectal Neoplasms; Lymph Nodes; Lymph Node Revealing Solution
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — methacarn; gewf solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colon Cancer (Active Comparator): The subjects in this group will undergo intervention by having surgery and lymph node clearing technique.
  Intervention A: Carnoy solution Intervention B: GEWF solution
  Interventions: Other: Lymph node clearing technique with Carnoy solution; Other: Lymph node clearing technique with GEWF solution
- Rectal Cancer (Active Comparator): The subjects in this group will undergo intervention by having surgery and lymph node clearing technique.
  Intervention A: Carnoy solution Intervention B: GEWF solution
  Interventions: Other: Lymph node clearing technique with Carnoy solution; Other: Lymph node clearing technique with GEWF solution

INTERVENTIONS:
Other: Lymph node clearing technique with Carnoy solution — Procedure: lymph node clearing technique with Carnoy solution
  (1) just after the surgical resection each specimen is fixed by formaldehyde; (2) lymph node harvesting is performed by a manual technique of vision and palpation; (3) lymph nodes retrieved are counted, stained with hematoxylin and eosin and examined with light microscopy; (4) the surgical specimen is submitted to re-fixation with Carnoy solution and another lymph node harvesting by manual technique of vision and palpation; (5) additional lymph nodes retrieved are counted, stained with hematoxylin and eosin and examined with light microscopy.
  Other Names: Carnoy
Other: Lymph node clearing technique with GEWF solution — Procedure: lymph node clearing technique with GEWF solution
  (1) just after the surgical resection each specimen is fixed by formaldehyde; (2) lymph node harvesting is performed by a manual technique of vision and palpation; (3) lymph nodes retrieved are counted, stained with hematoxylin and eosin and examined with light microscopy; (4) the surgical specimen is submitted to re-fixation with GEWF solution and another lymph node harvesting by manual technique of vision and palpation; (5) additional lymph nodes retrieved are counted, stained with hematoxylin and eosin and examined with light microscopy.
  Other Names: GEWF

SUMMARY:
Regional lymph node metastasis is a major determinant of local recurrence and overall survival rates in patients with colorectal cancer. Because of the poor prognosis associated with the presence of lymph node metastasis, stage III colorectal cancer patients should receive adjuvant treatment with chemo and / or radiation therapy according to the site of tumor. Several authors have investigated the use of revealing solutions for lymph node clearance in colorectal cancer. Most studies comparing conventional histopathological specimen examination to any lymph node clearing technique showed that the use of revealing solutions increases the mean number of lymph nodes harvested, usually in a statistically significant manner. It is still controversial the impact of the use of revealing solutions for upstaging of lymph node status and consequently for the indication for adjuvant therapy. Therefore will be conducted a randomized clinical trial to compares the performance of GEWF and Carnoy solutions for the histopathological examination of patients with colorectal cancer. The aim of this study is to determine the lymph node revealing solution with the best performance (increase in the mean number of lymph node harvested and lymph node upstaging) in patients with colorectal cancer.

DETAILED DESCRIPTION:
Patients with histologically proven colorectal adenocarcinoma submitted to curative resection and conventional histopathological examination of the surgical specimen are randomized to undergo further investigation by lymph node clearing technique with Carnoy or GEWF solution.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven colorectal adenocarcinoma
* Voluntary agreement of the patient to participate in research
* Voluntary agreement of the surgeon to participate in research

Exclusion Criteria:

* Absence of accurate histopathological data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-02 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Lymph nodes harvested | One week
  Number of additional lymph nodes harvested with the clearing technique

SECONDARY OUTCOMES:
Lymph node metastasis | One week
  Presence of metastasis in the additional lymph nodes harvested
Upstage of lymph nodes | One week
  Diagnosis of lymph node metastasis in a patient initially classified as having no lymph node metastasis or increase in the number of metastatic lymph nodes in a patient already staged as having lymph node metastasis.
Adjuvant therapy | One month
  Indication of adjuvant therapy as consequence of the upstaging after the lymph nodes clearing technique.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio N Kalil, MD, PhD, Principal Investigator — Researcher
Locations (1):
- Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul, Brazil